CLINICAL TRIAL: NCT04536558
Title: Olanzapine Plus Fosaprepitant Standard Antiemetic Therapy in the Prevention of Chemotherapy-induced Nausea and Vomiting in Patients Receiving High Emetic Risk Multi-day Chemotherapy: a Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 3 Study（OFFER）
Brief Title: Olanzapine Plus Fosaprepitant Standard Antiemetic Therapy in the Prevention of Chemotherapy-induced Nausea and Vomiting in Patients Receiving High Emetic Risk Multi-day Chemotherapy: a Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 3 Study
Acronym: OFFER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Li Zhang, MD, head of the medical department, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HS-TN-001
Record Dates: First submitted 2020-08-25; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Solid Tumor Patients Receiving High Emetic Risk Multi-day Chemotherapy
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- olanzapine plus fosaprepitant-based triple regimen (Experimental): Olanzapine（5mg p.o. d1-d5）plus fosaprepitant（150mg i.v. d1-d3） plus ondansetron（8mg i.v. d1-d3）and dexamethasone（6mg p.o. d1-d5） before undergoing chemotherapy.
  Interventions: Drug: olanzapine plus fosaprepitant-based triple regimen
- Placebo plus fosaprepitant-based triple regimen (Placebo Comparator): Placebo plus fosaprepitant（150mg i.v. d1-d3） plus ondansetron（8mg i.v. d1-d3）and dexamethasone（6mg p.o. d1-d5） before undergoing chemotherapy.
  Interventions: Drug: placebo plus fosaprepitant-based triple regimen

INTERVENTIONS:
Drug: olanzapine plus fosaprepitant-based triple regimen — olanzapine 5mg p.o. on day 1-day 5, fosaprepitant 150mg i.v. on day 1 before undergoing chemotherapy. Patients received ondansetron hydrochloride(8mg, i.v. day 1-day 3) and dexamethasone(6mg, oral, day 1-day 5) at the same time, before undergoing chemotherapy.
  Arms: olanzapine plus fosaprepitant-based triple regimen
Drug: placebo plus fosaprepitant-based triple regimen — placebo p.o. on day 1-day 5, fosaprepitant 150mg i.v. on day 1 before undergoing chemotherapy. Patients received ondansetron hydrochloride(8mg, i.v. day 1-day 3) and dexamethasone(6mg, oral, day 1-day 5) at the same time, before undergoing chemotherapy.
  Arms: Placebo plus fosaprepitant-based triple regimen

SUMMARY:
This is a multicenter, randomized, controlled, double-blind, phase III study.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, double-blind, phase III study assessing the efficacy and safety of Olanzapine plus fosaprepitant plus ondansetron and dexamethasone versus fosaprepitant plus ondansetron and dexamethasone in the prevention of chemotherapy-induced nausea and vomiting in patients receiving high emetic risk multi-day chemotherapy. Eligible patients will be randomized to receive either olanzapine plus fosaprepitant standard antiemetic therapy or fosaprepitant standard antiemetic therapy in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria: (abbreviated)

1. Male and female patients aged ≥ 18 and ≤ 75 years old;
2. Patients were diagnosed with histologically or cytology confirmed solid malignant tumors;
3. Patients have a Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2;
4. Patients were predicted life expectancy of ≥ 3 months;
5. Patients who were scheduled for 3 days of cisplatin based chemotherapy.

Exclusion Criteria: (abbreviated)

1. Patients were mentally disable or suffered from emotional disorders;
2. Patients were current illicit drug use, including alcohol abuse;
3. Patients scheduled administration of stem cell rescue therapy during cisplatin chemotherapy;
4. Patients have participated in other clinical trials in the past 4 weeks;
5. Patients were treated with chemotherapy including ordinary paclitaxel(using castor oil as a solvent);
6. Patients with active infections (e.g., pneumonia) or any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction) other than malignant tumors, and the researchers believe that it may confound the results of the study or expose patients receiving treatment with the study drug at unnecessary risk;
7. Patients have any disease that the researcher believes may confound the results of the study or expose the patient to unnecessary risk；
8. Patients were treated with moderate or highly emetogenic chemotherapy within 6 days prior to the initial of cisplatin infusion and/or 6 days after cisplatin infusion;
9. Patients were scheduled to receive radiation therapy to the abdomen or pelvis within a week of treatment;
10. Absolute neutrophil count<1,500 cells/ L, white blood cell count<3,000 cells/ L, platelet count<100,000 cells/ L, aspartate aminotransferase and alanine aminotransferase>2.5 upper limit of normal (ULN), bilirubin > 1.5 ULN, and creatinine > 1.5 ULN;
11. Patients were pregnant or breastfeeding;
12. Patients had suffered from vomiting or nausea in the 24 hours before treatment;
13. Patients were known to be at risk for narrow angle glaucoma；
14. Patients who are taking or have used CYP3A4 inducers within 30 days before the first day of treatment, which will affect the efficacy of the treatment drugs according to the researcher's evaluation, can not be enrolled;
15. Patients who are taking or have used CYP3A4 substrates and inhibitors within 7 days before the first day of treatment will significantly increase the treatment drug-related adverse events according to the researcher's evaluation, can not be enrolled;
16. Within 48 hours before the first day of treatment, patients used the following antiemetic agents: 5-hydroxytryptamine 3 receptor antagonists (such as ondansetron), phenothiazines (such as prochlorperazine), benzophenones (such as haloperidol), benzamide (such as metoclopramide), domperidone, cannabinoids, herbs with potential antiemetic effects, scopolamine, and cyclizine, etc;
17. Patients began to receive benzodiazepines or opioids within 48 hours prior to the first day of the study (except for triazolam, temazepam or midazolam single dose daily);
18. Patients had symptomatic primary or metastatic central nervous system malignancies;
19. Patients had concomitant diseases that could not take dexamethasone for 5 days, such as systemic fungal infection or uncontrolled diabetes mellitus;
20. Patients were not allowed to receive any dose of systemic glucocorticoid therapy within 72 hours before the first day except those prescribed in the protocol; however, local and inhaled corticosteroids were allowed;
21. Patients had a history of hypersensitivity to fosaprepitant meglumine, olanzapine, ondansetron or dexamethasone；
22. Patients had been treated with neurokinin-1 receptor antagonist in the past;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) during overall phase | Day 1 to day 8 after highly emetogenic chemotherapy initiation
  To compare olanzapine plus fosaprepitant regimen with placebo plus fosaprepitant regimen with respect to efficacy; complete response (CR) defined as no vomiting and no use of rescue therapy during overall phase (day 1 to day 8） after highly emetogenic chemotherapy initiation)

SECONDARY OUTCOMES:
Complete response (CR) during acute phase | Day 1 to day 3 days after highly emetogenic chemotherapy initiation
Complete response (CR) during delayed phase | Day 4 to day 8 after highly emetogenic chemotherapy initiation
No significant nausea during overall phase using questionnaire | Day 1 to day 8 after highly emetogenic chemotherapy initiation
No significant nausea during acute phase using questionnaire | Day 1 to day 3 after highly emetogenic chemotherapy initiation
No significant nausea during delayed phase using questionnaire | Day 4 to day 8 after highly emetogenic chemotherapy initiation
To compare quality of life using the functional living index-emesis questionnaire | From baseline to day 8 after highly emetogenic chemotherapy initiation
To compare olanzapine plus fosaprepitant regimen with placebo plus fosaprepitant regimen in terms of the number of days to first emetic episode. | Day 1 to day 8 after highly emetogenic chemotherapy initiation
To compare the number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From baseline to day 8 after highly emetogenic chemotherapy initiation
To compare the change of score using Hospital Anxiety and Depression Scale | From baseline to day 8 after highly emetogenic chemotherapy initiation
  Hospital Anxiety and Depression Scale includes two subscales: anxiety and depression, with 7 items for anxiety (a) and depression (d) respectively. Each item is divided into four grades of 0-3. The higher the score is, the more serious the anxiety and depression are.

OTHER OUTCOMES:
The plasma concentration of 5-hydroxytryptamine and substance P at the baseline | From baseline to day 8 after highly emetogenic chemotherapy initiation
  To explore the relationship between plasma concentration of 5-hydroxytryptamine、substance P and efficacy

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital& Institute, Chengdoucun
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Sun Yat-sen University Cancer Center, Guangdong
  - Harbin Medical University Cancer Hospital, Haerbin
  - Anhui Provincial Cancer Hospital, Hefei
  - Yunnan Cancer Hospital, Kunming
  - Jiangxi Cancer Hospital, Nanchang
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Fourth Hospital of Hebei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao Y, Yang Y, Gao F, Hu C, Zhong D, Lu M, Yuan Z, Zhao J, Miao J, Li Y, Zhu J, Wang C, Han J, Zhao Y, Huang Y, Zhang L. A multicenter, randomized, double-blind, placebo-controlled, phase 3 trial of olanzapine plus triple antiemetic regimen for the prevention of multiday highly emetogenic chemotherapy-induced nausea and vomiting (OFFER study). EClinicalMedicine. 2022 Dec 15;55:101771. doi: 10.1016/j.eclinm.2022.101771. eCollection 2023 Jan. PMID 36712888